CLINICAL TRIAL: NCT00597818
Title: A Multi-center, Randomized, Placebo-controlled, Double-blinded Study of the Efficacy and Safety of Cobiprostone for the Prevention of NSAID-induced Gastroduodenal Injury in Patients With Osteoarthritis and/or Rheumatoid Arthritis Patients
Brief Title: Cobiprostone Prevention of NSAID-induced Gastroduodenal Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU0621
Record Dates: First submitted 2008-01-10; First posted 2008-01-18 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2018-03

CONDITIONS: NSAID-induced Gastroduodenal Injury; Ulcers; Rheumatoid Arthritis; Osteoarthritis
MeSH Terms: conditions — Ulcer; Arthritis, Rheumatoid; Osteoarthritis | interventions — cobiprostone; Anti-Inflammatory Agents, Non-Steroidal; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants receive matching placebo capsules for 20 months
  Interventions: Drug: Placebo; Drug: Non-steroidal anti-inflammatory drug
- Cobiprostone QD (Experimental): Participants receive 18 mcg cobiprostone once daily (QD) for 20 months
  Interventions: Drug: Cobiprostone; Drug: Non-steroidal anti-inflammatory drug
- Cobiprostone BID (Experimental): Participants receive 18 mcg cobiprostone twice daily (BID) for 20 months
  Interventions: Drug: Cobiprostone; Drug: Non-steroidal anti-inflammatory drug
- Cobiprostone TID (Experimental): Participants receive 18 mcg cobiprostone three times daily (TID) for 20 months
  Interventions: Drug: Cobiprostone; Drug: Non-steroidal anti-inflammatory drug

INTERVENTIONS:
Drug: Cobiprostone — 18 mcg cobiprostone capsules for oral administration
  Other Names: SPI-8811; RU-8811
  Arms: Cobiprostone BID; Cobiprostone QD; Cobiprostone TID
Drug: Placebo — Matching placebo capsules for oral administration
  Other Names: Matching Placebo
  Arms: Placebo
Drug: Non-steroidal anti-inflammatory drug — Any marketed non-steroidal anti-inflammatory drug used by the participants as standard care.
  Other Names: Standard Care

SUMMARY:
The primary purpose of this study is to determine the efficacy and safety of three dose levels of cobiprostone as compared to placebo in OA/RA patients treated with an NSAID for 20 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient is more than 40 and less than 70 years of age.
* Patient has confirmed osteoarthritis (OA) and/or rheumatoid arthritis (RA) and could benefit from NSAID therapy.
* No current gastrointestinal H. pylori infection.

Exclusion Criteria:

* Known allergy or hypersensitivity to NSAIDs, or has any other contraindicated condition(s) to NSAID therapy.
* Patient has undergone a gastrointestinal or abdominal surgical procedure within 90 days prior to the Screening Visit, or has had a bowel resection at any time.
* Medical history includes prior or active GI complications and/or disorders, including but not limited to Barrett's esophagus, erosive esophagitis, esophageal stricture or ring, gastric obstruction, irritable bowel syndrome (IBS), or inflammatory bowel disease (IBD).
* Active symptomatic peptic ulcer disease or GI bleeding.
* Patient has received cobiprostone (SPI-8811; RU-8811) or AMITIZA (other names: lubiprostone, SPI-0211, or RU-0211) at any time prior to participation in this study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2007-08; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (19):
- United States (19):
  - Carl T Hayden VA Medical Center, Phoenix, Arizona
  - Gregory J. Wiener, MD PC, Chula Vista, California
  - Loma Linda University Physicians Medical Group, Loma Linda, California
  - Facey Medical Foundation, Mission Hills, California
  - Desert Oasis Healthcare, Palm Springs, California
  - Sepulveda Ambulatory Care Center, Sepulveda, California
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - University of Illinois Medical Center, Chicago, Illinois
  - Gulf Coast Research, LLC, Baton Rouge, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - Research Associates of New York, New York, New York
  - University of North Carolina Gastroenterology, Chapel Hill, North Carolina
  - Oklahoma Founddation for Digestive Research, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Gastroenterology Section at Temple University Hospital, Philadelphia, Pennsylvania
  - Dallas VA Research Corporation, Inc., Dallas, Texas
  - Houston Institute for Clinical Research, Houston, Texas
  - Digestive and Liver Disease Specialists, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 124 participants recruited, only 121 were actually enrolled.
Groups:
- Placebo: Matching placebo
- 18 mcg: Cobiprostone 18 mcg once daily (QD)
- 36 mcg: Cobiprostone 18 mcg twice daily (BID)
- 54 mcg: Cobiprostone 18 mcg three times daily (TID)
Period: Overall Study
Arm/Group | Placebo | 18 mcg | 36 mcg | 54 mcg
Started | 30 | 30 | 31 | 30
Completed | 12 | 14 | 12 | 20
Not Completed | 18 | 16 | 19 | 10

BASELINE CHARACTERISTICS:
Population: All subjects recruited were included in the baseline analysis set. Of the 124 participants recruited, only 121 were actually enrolled.
Groups:
- Cobiprostone QD: Cobiprostone 18 mcg once daily (QD)
- Cobiprostone BID: Cobiprostone 18 mcg twice daily (BID)
- Cobiprostone TID: Cobiprostone 18 mcg three times daily (TID)
- Total: Total of all reporting groups
Arm/Group | Placebo | Cobiprostone QD | Cobiprostone BID | Cobiprostone TID | Total
Number analyzed (Participants) | 32 | 30 | 31 | 31 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 27 | 27 | 29 | 112
  >=65 years | 3 | 3 | 4 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (7.9) | 53.9 (8.01) | 54.6 (8.28) | 53.3 (8.18) | 54.0 (8.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 23 | 24 | 90
  Male | 9 | 10 | 8 | 7 | 34
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 30 | 31 | 31 | 124

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Gastric Ulcers
Time Frame: at 20 months
Population: Intention to treat (ITT) population, defined as all participants enrolled in the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cobiprostone QD | Cobiprostone BID | Cobiprostone TID
Number analyzed (Participants) | 30 | 30 | 31 | 30
Participants | 7 | 5 | 7 | 4

2. Secondary Outcome: Number of Participants With Duodenal and Gastroduodenal Ulcers
Time Frame: at 20 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cobiprostone QD | Cobiprostone BID | Cobiprostone TID
Number analyzed (Participants) | 30 | 30 | 31 | 30
Participants | 1 | 4 | 1 | 2

3. Secondary Outcome: Number of Participants With Gastric, Duodenal, and Gastroduodenal Ulcers
Time Frame: at Week 4
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cobiprostone QD | Cobiprostone BID | Cobiprostone TID
Number analyzed (Participants) | 30 | 30 | 31 | 30
Participants | 7 | 8 | 8 | 6

4. Secondary Outcome: Size of Ulcers/Erosions
Time Frame: at 20 Months
Population: ITT
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Cobiprostone QD | Cobiprostone BID | Cobiprostone TID
Number analyzed (Participants) | 30 | 30 | 31 | 30
mm | 8.5 (20.49) | 4.7 (2.63) | 3.5 (2.35) | 2.6 (1.54)

ADVERSE EVENTS:
Time Frame: All participants were treated and followed for ulcers and other adverse events for a total of 20 months
Arm/Group | Placebo | Cobiprostone QD | Cobiprostone BID | Cobiprostone TID
Serious Adverse Events (participants affected / at risk) | 22/30 | 23/30 | 25/31 | 26/30
Other Adverse Events (participants affected / at risk) | 20/30 | 18/30 | 22/31 | 21/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Cobiprostone QD (N=30) | Cobiprostone BID (N=31) | Cobiprostone TID (N=30)
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 11 | 12
Nausea (Gastrointestinal disorders) | 4 | 3 | 5 | 5
Dyspepsia (Gastrointestinal disorders) | 6 | 3 | 2 | 5
Gastritis (Gastrointestinal disorders) | 5 | 4 | 2 | 3
Erosive oesophagitis (Gastrointestinal disorders) | 6 | 3 | 2 | 2
Flatulence (Gastrointestinal disorders) | 4 | 4 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 3 | 2
Duodenitis (Gastrointestinal disorders) | 3 | 3 | 1 | 3
Hiatus hernia (Gastrointestinal disorders) | 0 | 3 | 2 | 3
Gastrointestinal tract mucosal discolouration (Gastrointestinal disorders) | 2 | 3 | 1 | 2
Reflux oesophagitis (Gastrointestinal disorders) | 3 | 3 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 3 | 2 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Cobiprostone QD (N=30) | Cobiprostone BID (N=31) | Cobiprostone TID (N=30)
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 10 | 11
Nausea (Gastrointestinal disorders) | 3 | 3 | 5 | 5
Dyspepsia (Gastrointestinal disorders) | 5 | 2 | 1 | 4
Gastritis (Gastrointestinal disorders) | 4 | 4 | 2 | 3
Erosive Oesophagitis (Gastrointestinal disorders) | 5 | 2 | 2 | 2
Flatulence (Gastrointestinal disorders) | 4 | 3 | 1 | 2
Abdominal Pain Other (Gastrointestinal disorders) | 3 | 2 | 3 | 2
Duodenitis (Gastrointestinal disorders) | 3 | 3 | 1 | 3
Reflux oesphagitis (Gastrointestinal disorders) | 3 | 2 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 3 | 2 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Oesophagitis (Gastrointestinal disorders) | 2 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other